CLINICAL TRIAL: NCT03614403
Title: The Effect of Single High Dose of Vitamin D3 on Short-term Postoperative Pain in Patients Under Craniotomy for Brain Tumor Resection
Brief Title: The Effect of Vitamin D3 on Postoperative Pain in Patients Undergoing Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1397.271
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Intervention patients will be received a single dose of 300000 IU vitamin D via intramuscular injection
  Interventions: Drug: vitamin D
- control (No Intervention): Control patients will not be received any intervention

INTERVENTIONS:
Drug: vitamin D — Fat-soluble vitamin D injection contain of 300,000 IU vitamin D that given via intramuscular injection
  Other Names: Cholecalciferol
  Arms: Vitamin D

SUMMARY:
Vitamin D is a hormone mainly synthesized in the skin in the presence of sunlight. Like other hormones, vitamin D plays a role in a wide range of processes in the body. Some studies have shown vitamin D has anti-inflammatory effects in the body by reducing the release of pro-inflammatory cytokines and suppressing T-cell responses. Therefore, vitamin D may be effective on reduce pain by such mechanisms. In this trial patients with brain tumor under craniotomy will receive a single high dose vitamin D compared to the control group.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in intensive care unit (ICU) and neurosurgery ward, in Shohada-E-Tajrish hospital,Tehran, Iran. First, patients will be carefully checked for inclusion and exclusion criteria. Then, the eligible patients will complete the consent form for this study. 60 eligible brain tumor patients diagnosed by surgeon that are ready for craniotomy will be selected.These patients will be divided into two groups. Intervention group will be received an intramuscular (IM) single dose of vitamin D (300000 IU),while another group will not receive. Pain in patients will be checked daily by up to 3 days after surgery. Finally, the VAS pain score will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of patient or legal representative
* 25(OH)D level below 20ng/dL

Exclusion Criteria:

* Other trial participation, including previous participation in the pilot trial
* Pregnant or lactating women
* Hypercalcemia
* Hyperphosphatemia
* Tuberculosis
* Sarcoidosis
* History of nephrolithiasis
* History of hyperparathyroidism
* Medications that interfere with vitamin D metabolism
* Renal Insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Short-term postoperative pain: measured by the visual analogue scale or visual analog scale (VAS) that is a pain rating scale | Up to three days after surgery
  By questioning from patients for daily pain intensity based on the VAS scale in which pain intensity score by 0 to 10. The "0" and "10" score indicates "no pain" and "worst pain",respectively. also "1-3" , "4-6" and "7-9" score indicates mild, mild to moderate and severe pain, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, PhD, Study Chair — Faculty of Nutrition and Food Technology,
Locations (1):
- Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No